CLINICAL TRIAL: NCT05909735
Title: Treatment of Limbal Stem Cell Deficiency With Descemet's Membrane
Brief Title: Treatment of LSCD With DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPH-2023-31727
Record Dates: First submitted 2023-03-29; First posted 2023-06-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Limbal Stem-cell Deficiency; Congenital Aniridia
Keywords: congenital aniridia; limbal stem cell deficiency; Descemet's Membrane
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Aniridia

STUDY DESIGN:
Intervention Model Description: This is an interventional non-comparative pilot clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visually significant partial LSCD (Experimental): Patient with visually significant partial LSCD, as defined by a best corrected visual acuity of 20/100 or less, and partial LSCD on slit lamp exam with at least 25% of the limbus intact or at least 25% of the corneal surface covered with corneal epithelium will be enrolled in the first arm.
  Interventions: Procedure: transplantation of a Descemet's Membrane corneal onlay, partial LSCD
- Total/near-total LSCD with recurrent or persistent epithelial defects (PED) (Experimental): Patient with visually significant total LSCD, as defined by a best corrected visual acuity of 20/100 or less, and total LSCD on slit lamp exam with over 25% of the limbus intact or less than 25% of the corneal surface covered with corneal epithelium; and a history of a persistent epithelial defect that has persisted over 2 weeks despite maximal medical therapy, or a history of recurrent epithelial erosions that occur more frequently than once a month; will be enrolled in the second arm.
  Interventions: Procedure: transplantation of a Descemet's Membrane corneal onlay, total/near-total LSCD

INTERVENTIONS:
Procedure: transplantation of a Descemet's Membrane corneal onlay, partial LSCD — The worst seeing eye of these patients (or a randomized eye if vision is equal bilaterally) will be treated with superficial keratectomy to remove any pannus and debride the central corneal epithelium, followed by transplantation of a Descemet's membrane corneal onlay. Patient will be followed for 6 months and evaluated for improvement in visual acuity and improvement in limbal stem cell deficiency, and monitored for adverse events.
  Arms: Visually significant partial LSCD
Procedure: transplantation of a Descemet's Membrane corneal onlay, total/near-total LSCD — The worst seeing eye of these patients (or a randomized eye if vision is equal bilaterally) will be treated with superficial keratectomy to remove any pannus and debride the central corneal epithelium, followed by transplantation of a Descemet's membrane (DM) corneal onlay. Patient will be followed for 6 months and evaluated for improvement in visual acuity, limbal stem cell deficiency, and persistent epithelial defects/recurrent erosions, and monitored for adverse events.
  Arms: Total/near-total LSCD with recurrent or persistent epithelial defects (PED)

SUMMARY:
Limbal Stem Cell Deficiency (LSCD) is a blinding disease that accounts for an estimated 15-20% of corneal blindness worldwide. Current treatments are limited. Traditional corneal transplantation with penetrating keratoplasty (PKP) is ineffective in treating these patients. Without a healthy population of limbal stem cells (LSC) to regenerate the corneal epithelium, standard corneal transplants will not re-epithelialize and will rapidly scar over or melt.

The limbal niche is the microenvironment surrounding the LSCs that is critical for maintaining their survival and proliferative potential under physiologic conditions. Extracellular signals from the microenvironment are critical to the normal function and maintenance of pluripotent stem cells. Identifying an effective niche replacement is thus an important focus of limbal stem cell research and critical for advancing treatments for LSCD.

Descemet's membrane (DM), an acellular, naturally occurring, basement membrane found on the posterior surface of the cornea, is a promising niche replacement. DM is routinely isolated and transplanted intraocularly with associated donor corneal endothelium for treatment of diseases like Fuchs' dystrophy and corneal bullous keratopathy that specifically affect DM and corneal endothelium. However, its application on the ocular surface has not been explored. DM is optically clear and highly resistant to collagenase digestion. This makes it very attractive as a long-term corneal on-lay and niche replacement on the surface of the eye. The anterior fetal banded layer of DM shares key compositional similarities with limbal basement membrane, which is a major component of the limbal niche. These similarities include limbus-specific extracellular matrix proteins such as collagen IV that is restricted to the α1, α2 subtypes, vitronectin, and BM40/SPARC. Of these, vitronectin and BM40/SPARC are known to promote proliferation of LSCs and induced pluripotent stem cells (iPSC) in culture.

Because of this, DM is a promising biological membrane for establishing a niche-like substrate on the corneal surface in patients with LSCD. The purpose of this pilot study is to investigate the clinical efficacy of using DM as a corneal on-lay to promote corneal re-epithelialization in partial LSCD.

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* partial LSCD (involving less than 75% of the limbus, or <75% of the corneal surface)
* Visually significant (best-corrected visually acuity 20/100 or worse)

Arm 2:

* total/near-total LSCD with recurrent erosions or PEDs (involving more than 75% of the limbus, or more than 75% of the corneal surface)
* Visually significant (best-corrected visually acuity 20/100 or worse) PLUS
* Persistent epithelial defects last >2 weeks despite maximal medical therapy OR
* Recurrent erosions occuring at least once every month

Exclusion Criteria:

* Pregnant women
* Prisoners (vulnerable population)
* Adults lacking capacity to consent (vulnerable population)
* Adults unable to sign consent due to non-english speaking or illiterate (vulnerable population)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Visual improvement | 180 days following intervention
  Visual Acuity: Improvement in visual acuity over time will be measured as the difference in post-op visual acuity at post-operative week 1, month 1, month 3, and month 6 compared to pre-op visual acuity. Visual acuity will be assessed in study eyes with a standard Snellen Eye Chart.
Graft Retention on Slit Lamp Examination | 180 days following intervention
  Retention of the graft: Retention of the graft on the surface of the eye will be documented as present, absent, or indeterminant using slit lamp examination. For slit lamp examination, retention of the graft will be evidenced by visualization of a gentian violet orientation mark (s-stamp) that will be placed on all grafts at the time of tissue processing by the eye bank (prior to transplantation).
Graft Retention on Slit Lamp Photography. | 180 days following intervention
  Retention of the graft: In order to maintain photographic proof of the findings on slit lamp examination, slit lamp photography will also be taken. Study eyes will be photographed at the slit lamp at post-operative week 1, month 1, month 3, and month 6. Retention of the graft will be evidenced by visualization of a gentian violet orientation mark (s-stamp) that will be placed on all grafts at the time of tissue processing by the eye bank (prior to transplantation). This photographic documentation will assist in confirming the findings in outcome measure #2.
Incidence of Post-operative Adverse Events Requiring Treatment | 180 days following intervention
  Post-operative adverse events: Patients will be assessed at slit lamp at post-operative week 1, month 1, month 3, and month 6 for dislocation or opacification of the DM corneal onlay, PEDs, elevated intraocular pressure (IOP), and/or infectious keratitis to assess the safety of the therapy. Any persistent epithelial defect will be measured for size on slit lamp by recording the long and short diameter of any defect. IOP will be measured using a Goldman applanation. Infectious keratitis and membrane dislocation will be assessed at slit lamp during each post-operative visit.
Corneal Neovascularization on Slit Lamp Examination | 180 days following intervention
  Corneal Neovascularization: will be evaluated using slit lamp examination pre-operatively and post-operatively at week 1, month 1, month 3, and month 6. The degree of corneal neovascularization will be quantified using a previously established 10-point slit lamp examination score based on the extent of limbal involvement (number of quadrants involved - up to 4 points), the extent of corneal surface involvement (total area of corneal involved - up to 4 points), and whether the central visual axis is involved (up to 2 points).
Corneal Neovascularization on Slit Lamp Photography | 180 days following intervention
  In order to maintain photographic proof of the findings on slit lamp examination, slit lamp photography will also be taken. Photos will be taken pre-operatively and post-operatively at week 1, month 1, month 3, and month 6. The degree of corneal neovascularization on the photos will be compared to the documented 10-point slit lamp examination score from outcomes measure #6 to confirm the accuracy of the results. Again, the 10-point slit lamp examination score is based on the extent of limbal involvement (number of quadrants involved - up to 4 points), the extent of corneal surface involvement (total area of corneal involved - up to 4 points), and whether the central visual axis is involved (up to 2 points).
Corneal Epitheliopathy on Slit Lamp Examination | 180 days following intervention
  Corneal Epitheliopathy: will be evaluated using slit lamp examination pre-operatively and post-operatively at week 1, month 1, month 3, and month 6. The degree of corneal epitheliopathy will be quantified using a previously established 10-point slit lamp examination score based on the extent of limbal involvement (number of quadrants involved - up to 4 points), the extent of corneal surface involvement (total area of corneal involved - up to 4 points), and whether the central visual axis is involved (up to 2 points).
Corneal Epitheliopathy on Slit Lamp Photography | 180 days following intervention
  In order to maintain photographic proof of the findings on slit lamp examination, slit lamp photography will also be taken. Photos will be taken pre-operatively and post-operatively at week 1, month 1, month 3, and month 6. The degree of corneal epitheliopathy on the photos will be compared to the documented 10-point slit lamp examination score from outcomes measure #8 to confirm the accuracy of the results. Again, the 10-point slit lamp examination score is based on the extent of limbal involvement (number of quadrants involved - up to 4 points), the extent of corneal surface involvement (total area of corneal involved - up to 4 points), and whether the central visual axis is involved (up to 2 points).
Corneal epithelial thickness | 180 days following intervention
  Corneal epithelial thickness will be assessed as a metric of LSCD severity. Corneal epithelial thickness will be measured in cross-section on AS-OCT only.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kaufman, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States